CLINICAL TRIAL: NCT00625482
Title: Sex-Differential Health Interventions In Low-Birth-Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: March of Dimes (Other); Danida (Unknown)
Purpose: Prevention
Other Study IDs: 2007-7041-121
Record Dates: First submitted 2008-02-18; First posted 2008-02-28 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Mortality; Morbidity; Growth; Neonatal Mortality
Keywords: BCG vaccine; Oral polio vaccine; Vitamin A supplementation; Low-birth-weigth; Sex-differential; Prevention; Immunological parameters
MeSH Terms: interventions — Poliovirus Vaccine, Oral

ARMS (4):
- Boys 1 (Active Comparator): OPV as usual
  Interventions: Biological: OPV
- Boys 2 (Experimental): OPV plus BCG
  Interventions: Biological: OPV plus BCG
- Girls 1 (Active Comparator): OPV as usual
  Interventions: Biological: OPV
- Girls 2 (Experimental): OPV plus BCG
  Interventions: Biological: OPV plus BCG

INTERVENTIONS:
Biological: OPV
  Arms: Boys 1
Biological: OPV plus BCG
  Arms: Boys 2
Biological: OPV
  Arms: Girls 1
Biological: OPV plus BCG
  Arms: Girls 2

SUMMARY:
Our group has consistently found that the major interventions to reduce morbidity and mortality in low-income countries have sex-differential effects. These interventions include BCG vaccine, oral polio vaccination (OPV), and vitamin A supplementation (VAS).

Low-birth-weight (LBW) children constitute the largest high-risk group in low-income countries. According to current policy, they receive OPV at birth. Current evidence suggests that a policy of providing BCG with OPV for girls and VAS instead of OPV for boys at birth may improve survival in LBW neonates. This will be tested in a large randomized trial.

We experienced an unexpected cluster of deaths among boys in the VAS arm, which could be due to chance, but we decided to stop randomizing boys to OPV or VAS. Very recent evidence has suggested that low-birth-weight boys may benefit from BCG at birth as well. Hence, we have obtained ethical permission to continue the trial with randomization of boys to OPV or OPV plus BCG.

ELIGIBILITY:
Inclusion Criteria:

* Low-birth-weight infants (<2500 g)

Exclusion Criteria:

* Already received BCG/OPV
* Overtly sick or have malformations at the time of enrolment
* Clinical signs of vitamin A deficiency (very unlikely)

Max Age: 1 Month | Sex: All
Age Groups: Child
Dates: Start 2008-02

PRIMARY OUTCOMES:
Mortality

SECONDARY OUTCOMES:
Overall severe morbidity as measured by number of hospitalizations
Morbidity due to rotavirus and malaria
Growth
BCG scar formation and PPD delayed type hypersensitivity (DTH) response
Changes in cytokine profile

CONTACTS AND LOCATIONS:
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

REFERENCES:
- [Derived] Schaltz-Buchholzer F, Berendsen M, Roth A, Jensen KJ, Bjerregaard-Andersen M, Kjaer Sorensen M, Monteiro I, Aaby P, Stabell Benn C. BCG skin reactions by 2 months of age are associated with better survival in infancy: a prospective observational study from Guinea-Bissau. BMJ Glob Health. 2020 Sep;5(9):e002993. doi: 10.1136/bmjgh-2020-002993. PMID 32978212
- [Derived] Jensen KJ, Biering-Sorensen S, Ursing J, Kofoed PL, Aaby P, Benn CS. Seasonal variation in the non-specific effects of BCG vaccination on neonatal mortality: three randomised controlled trials in Guinea-Bissau. BMJ Glob Health. 2020 Mar 5;5(3):e001873. doi: 10.1136/bmjgh-2019-001873. eCollection 2020. PMID 32201619
- [Derived] Schaltz-Buchholzer F, Biering-Sorensen S, Lund N, Monteiro I, Umbasse P, Fisker AB, Andersen A, Rodrigues A, Aaby P, Benn CS. Early BCG Vaccination, Hospitalizations, and Hospital Deaths: Analysis of a Secondary Outcome in 3 Randomized Trials from Guinea-Bissau. J Infect Dis. 2019 Jan 29;219(4):624-632. doi: 10.1093/infdis/jiy544. PMID 30239767
- [Derived] Biering-Sorensen S, Aaby P, Lund N, Monteiro I, Jensen KJ, Eriksen HB, Schaltz-Buchholzer F, Jorgensen ASP, Rodrigues A, Fisker AB, Benn CS. Early BCG-Denmark and Neonatal Mortality Among Infants Weighing <2500 g: A Randomized Controlled Trial. Clin Infect Dis. 2017 Oct 1;65(7):1183-1190. doi: 10.1093/cid/cix525. PMID 29579158
- [Derived] Biering-Sorensen S, Jensen KJ, Monterio I, Ravn H, Aaby P, Benn CS. Rapid Protective Effects of Early BCG on Neonatal Mortality Among Low Birth Weight Boys: Observations From Randomized Trials. J Infect Dis. 2018 Feb 14;217(5):759-766. doi: 10.1093/infdis/jix612. PMID 29216358
- [Derived] Biering-Sorensen S, Jensen KJ, Aamand SH, Blok B, Andersen A, Monteiro I, Netea MG, Aaby P, Benn CS, Haslov KR. Variation of growth in the production of the BCG vaccine and the association with the immune response. An observational study within a randomised trial. Vaccine. 2015 Apr 21;33(17):2056-65. doi: 10.1016/j.vaccine.2015.02.056. Epub 2015 Mar 10. PMID 25765965
- [Derived] Lund N, Biering-Sorensen S, Andersen A, Monteiro I, Camala L, Jorgensen MJ, Aaby P, Benn CS. Neonatal vitamin A supplementation associated with a cluster of deaths and poor early growth in a randomised trial among low-birth-weight boys of vitamin A versus oral polio vaccine at birth. BMC Pediatr. 2014 Aug 28;14:214. doi: 10.1186/1471-2431-14-214. PMID 25163399
- [Derived] Eriksen HB, Biering-Sorensen S, Lund N, Correia C, Rodrigues A, Andersen A, Ravn H, Aaby P, Jeppesen DL, Benn CS. Factors associated with thymic size at birth among low and normal birth-weight infants. J Pediatr. 2014 Oct;165(4):713-21. doi: 10.1016/j.jpeds.2014.06.051. Epub 2014 Jul 30. PMID 25085521